CLINICAL TRIAL: NCT03658941
Title: Prophylactic Use of Dural Tenting Sutures in Elective Craniotomies - is it Necessary? A Multicentre Randomised Study.
Brief Title: Dural Tenting Sutures in Neurosurgery - is it Necessary?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KB/106/2018
Record Dates: First submitted 2018-08-31; First posted 2018-09-06 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2019-01

CONDITIONS: Epidural Hematoma
Keywords: craniotomy; dural tenting suture; epidural hematoma
MeSH Terms: conditions — Hematoma, Epidural, Spinal

STUDY DESIGN:
Intervention Model Description: We plan to include 2000 subjects in this study. Each subject will undergo a craniotomy for unrelated pathology. Each of the subjects will be assigned in random order to an intervention or control group. The intervention group will not have dural tenting sutures during closure of their craniotomy while the control group will have at least three.
  Both groups will be followed radiologically and clinically, in the exact same manner.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Due to the nature of the surgical procedures, the surgeon and the rest of the OR medical team will be aware of the current subject's allocation. However, in each case, the specific OR team aware of the subject's allocation will be different from the investigators performing further evaluation of the given subject. The following study procedures will be in place to ensure double-blind administration of the study.
  * Access to the randomization code will be strictly controlled.
  * The surgeon will receive information on subject's allocation after commencing the surgery.
  The study blind will be broken:
  1. During interim monitoring, after recruiting the first 100 patients.
  2. On completion of the clinical study and after the study database has been locked.
  3. When patients' safety requires access to allocation data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No dural tenting sutures (Experimental): No dural tenting techniques
  Interventions: Procedure: No dural tenting techniques
- Dural tenting sutures (Active Comparator): Dural tenting techniques
  Interventions: Procedure: Dural tenting techniques

INTERVENTIONS:
Procedure: No dural tenting techniques — Not applying dural tenting sutures during closure of a craniotomy
  Other Names: tack-up sutures; hitch-up stitches
  Arms: No dural tenting sutures
Procedure: Dural tenting techniques — Applying at least 3 dural tenting sutures during closure of a craniotomy
  Other Names: tack-up sutures; hitch-up stitches
  Arms: Dural tenting sutures

SUMMARY:
This study evaluates the necessity of dural tenting sutures in craniotomies. The sutures elevate the dura, a layer between the brain and skull. Supposedly, by doing so, they prevent blood collecting between dura mater and the skull. These blood collections, called epidural hematomas, contributed greatly to postoperative mortality in the early days of neurosurgery. There have been several reports questioning the ongoing need for them in neurosurgery, thanks to modern hemostatic techniques. Moreover, it has been published in the literature, and is a common knowledge as well, that some neurosurgeons do not use these sutures at all, and do not have worse outcomes than their colleagues.

In this study, half of the randomly assigned participants will undergo craniotomy without dural tenting sutures and will be considered an intervention group. The other half will undergo craniotomy with these sutures.

DETAILED DESCRIPTION:
In the early days of neurosurgery, epidural hemorrhages (EDH) contributed to a high mortality rate after craniotomies. Almost a century ago Walter Dandy reported dural tenting sutures as an effective way of preventing postoperative EDH. Over time, his technique gained in popularity and significance to finally become a neurosurgical standard.

Yet, there have been several retrospective reports questioning the ongoing need for dural tenting sutures. Dandy's explanation that the hemostasis under hypotensive conditions is deceiving and eventually causes EDH may be obsolete. These days, proper intra- and postoperative care, including maintenance of normovolemia and normotension and the use of modern hemostatic agents, may be enough for effective hemostasis. Evading of this suturing technique by some surgeons supports this argument even further.

Thus, there is a fundamental need to evaluate the necessity of dural tenting sutures in an unbiased, evidence-based manner.

ELIGIBILITY:
Inclusion Criteria:

* male or female over 18 and under 75 years old
* qualified for an elective supratentorial craniotomy with a diameter of at least 3 cm
* Glasgow Coma Scale 15 preoperatively
* Modified Rankin Scale 0, 1 or 2 preoperatively

Exclusion Criteria:

* Coagulation abnormalities before the surgery
* Revision craniotomy
* Skull base surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Reoperation due to epidural hematoma | During hospitalization for the surgery, approximately 2 days postoperatively
  Surgery for the postoperative extradural hematoma

SECONDARY OUTCOMES:
Postoperative 30-day mortality | 30-day postoperatively
  The data to measure postoperative 30-day mortality will be obtained from a national database 30 days after the recruitment of all participants has been completed.
Postoperative 30-day readmission to a neurosurgical or neurological department | 30-day postoperatively
  The data required to evaluate readmission rates will be obtained from the hospital databases.
New neurologic deficit or deterioration of a previous one | during hospitalisation, as evaluated 5-7 days postoperatively, or earlier if the patient is discharged before the fifth postsurgical day.
  New neurologic deficit or deterioration of a preoperative deficit, as evaluated on postoperative day 5-7.
Cerebrospinal fluid leak requiring treatment. | during hospitalisation, as evaluated 5-7 days postoperatively, or earlier if the patient is discharged before the fifth postsurgical day.
  Presence of a cerebrospinal fluid leak requiring treatment.
Deterioration of postoperative headaches over 5 Numerical Rating Scale | during hospitalisation, as evaluated 5-7 days postoperatively, or earlier if the patient is discharged before the fifth postsurgical day.
  The Numeric Rating Scale is an 11-point scale for patient self-reporting of pain. It ranges from 0 (no pain) to 10 (the worst imaginable pain). There are no subscales. Higher values indicate more pain and, therefore, represent undesirable outcome.
Epidural collection thickness over 3 mm measured radiographically | During hospitalization, approximately 1-3 days postoperatively
  Extradural collection thickness measured in postoperative Computed Tomography by two independent radiologists
Midline shift over 5 mm | During hospitalization, approximately 1-3 days postoperatively
  Extradural collection thickness measured in postoperative Computed Tomography by two independent radiologists

CONTACTS AND LOCATIONS:
Overall Officials: Łukasz Przepiórka, Principal Investigator — Department of Neurosurgery, Medical University of Warsaw; Przemysław Kunert, MD, PhD, Principal Investigator — Department of Neurosurgery, Medical University of Warsaw
Locations (5):
- Poland (5):
  - Department of Neurosurgery, 10th Military Research Hospital and Polyclinic, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - 5 Neurosurgery and Pediatric Neurosurgery Department in Lublin, Medical University of Lublin, Lublin, Lublin Voivodeship
  - Department of Neurosurgery, Medical University of Warsaw, Warsaw, Mazovian
  - Department of Neurosurgery, Medical University of Silesia, Regional Hospital, Sosnowiec, Sosnowiec, Silesian Voivodeship
  - Department of Neurosurgery and Oncology of Central Nervous System, Barlicki University Hospital, Medical University of Lodz, Lodz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: Undecided
The trial protocol, full study report, anonymised participant-level dataset and statistical code for generating the results will be made publicly available if all investigators agree to share the data.

REFERENCES:
- [Background] Swayne OB, Horner BM, Dorward NL. The hitch stitch: an obsolete neurosurgical technique? Br J Neurosurg. 2002 Dec;16(6):541-4; discussion 544. PMID 12617233
- [Background] Winston KR. Efficacy of dural tenting sutures. J Neurosurg. 1999 Aug;91(2):180-4. doi: 10.3171/jns.1999.91.2.0180. PMID 10433304
- [Background] Winston KR. Dural tenting sutures in pediatric neurosurgery. Pediatr Neurosurg. 1998 May;28(5):230-5. doi: 10.1159/000028656. PMID 9732254
- [Background] Wadanamby, S. et al., (2016). Is dural hitching necessary to prevent post-operative extradural haemorrhage in craniotomies and craniectomies. Sri Lanka Journal of Surgery. 34(2), pp.11-17. DOI: http://doi.org/10.4038/sljs.v34i2.8262
- [Derived] Przepiorka L, Wojtowicz K, Kujawski S, Wisniewski K, Bobeff EJ, Kruk R, Kulesza B, Fortuniak J, Mroz A, Dunaj P, Kaspera M, Hoppe S, Krystkiewicz K, Kwiecien K, Szczepanek D, Jaskolski DJ, Ladzinski P, Rola R, Furtak J, Trojanowski T, Marchel A, Kunert P. Dural Tenting in Elective Craniotomies: A Randomized Clinical Trial. Neurosurgery. 2025 Nov 1;97(5):1108-1117. doi: 10.1227/neu.0000000000003480. Epub 2025 May 1. PMID 40310111
- [Derived] Kunert P, Przepiorka L, Fortuniak J, Wisniewski K, Bobeff EJ, Larysz P, Kruk R, Kulesza B, Szczepanek D, Ladzinski P, Zylkowski J, Kujawski S, Labedzka K, Jaskolski D, Rola R, Trojanowski T, Marchel A. Prophylactic use of dural tenting sutures in elective craniotomies in adults-is it necessary? A study protocol for a multicentre, investigator- and participant-blinded randomised, parallel-group, non-inferiority trial. Trials. 2021 Apr 12;22(1):273. doi: 10.1186/s13063-021-05201-z. PMID 33845888
- See also: Website of the clinical trial — http://rctszwydandy.wum.edu.pl/en

DOCUMENTS (2):
  • Study Protocol (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT03658941/Prot_007.pdf
  • Statistical Analysis Plan (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT03658941/SAP_006.pdf